CLINICAL TRIAL: NCT01372085
Title: A Single Ascending Dose and Relative Bioavailability Study of LY2584702 in Healthy Subjects
Brief Title: Single Dose Study in Healthy Participants to Investigate the Safety and Absorption of LY2584702
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 14318; I3G-FW-JGCE (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-06-02; First posted 2011-06-13 (Estimated); Results first posted 2019-01-22 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2018-08

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Part A: 25 mg RF (Experimental): A single 25 mg dose of LY2584702 RF
  Interventions: Drug: LY2584702 Reference Formulation
- Part A: Placebo (Placebo Comparator): Placebo taken orally
  Interventions: Drug: Placebo
- Part B: Sequence 1 (Experimental): A single 10 mg dose of LY2584702 TF during the first intervention period, followed by placebo in the second intervention period, followed by a single dose of 50 mg TF in the third intervention period, followed by either an open-label single dose of 50 mg TF after a high fat breakfast (Period 4a) OR placebo or escalated dose of TF in the fasted state (Period 4b). There will be a washout period of at least 3 days between periods.
  Interventions: Drug: LY2584702 Test Formulation; Drug: Placebo
- Part B: Sequence 2 (Experimental): Placebo during the first intervention period, followed by a single dose of 50 mg RF in the second intervention period, followed by a single dose of 50 mg TF in the third intervention period, followed by either an open-label single dose of 50 mg TF after a high fat breakfast (Period 4a) OR placebo or escalated dose of TF in the fasted state (Period 4b). There will be a washout period of at least 3 days between periods.
  Interventions: Drug: LY2584702 Reference Formulation; Drug: LY2584702 Test Formulation; Drug: Placebo
- Part B: Sequence 3 (Experimental): A single 10 mg dose of LY2584702 TF during the first intervention period, followed by a single dose of 50 mg RF in the second intervention period, followed by a single dose of 50 mg TF in the third intervention period, followed by either an open-label single dose of 50 mg TF after a high fat breakfast (Period 4a) OR placebo or escalated dose of TF in the fasted state (Period 4b). There will be a washout period of at least 3 days between periods.
  Interventions: Drug: LY2584702 Reference Formulation; Drug: LY2584702 Test Formulation; Drug: Placebo
- Part B: Sequence 4 (Experimental): A single 10 mg dose of LY2584702 TF during the first intervention period, followed by a single dose of 50 mg RF in the second intervention period, followed by placebo in the third intervention period, followed by either an open-label single dose of 50 mg TF after a high fat breakfast (Period 4a) OR placebo or escalated dose of TF in the fasted state (Period 4b). There will be a washout period of at least 3 days between periods.
  Interventions: Drug: LY2584702 Reference Formulation; Drug: LY2584702 Test Formulation; Drug: Placebo

INTERVENTIONS:
Drug: LY2584702 Reference Formulation — Administered orally
  Arms: Part A: 25 mg RF; Part B: Sequence 2; Part B: Sequence 3; Part B: Sequence 4
Drug: LY2584702 Test Formulation — Administered orally
  Arms: Part B: Sequence 1; Part B: Sequence 2; Part B: Sequence 3; Part B: Sequence 4
Drug: Placebo — Administered orally
  Arms: Part A: Placebo; Part B: Sequence 1; Part B: Sequence 2; Part B: Sequence 3; Part B: Sequence 4

SUMMARY:
This is a single-centre, placebo-controlled, two-part study in healthy participants.

Part A will be a single dose, single period, placebo-controlled pilot study to explore the safety, tolerability, absorption and pharmacodynamic [effect of drug on a biological marker-phospho-S6 (pS6) levels in skin biopsies] of a single dose of 25 milligrams (mg) LY2584702 Reference formulation (RF). Part B is a single dose, placebo-controlled, 4-period crossover study to primarily evaluate the absorption of the Test Formulation (TF) in comparison with the (RF) of LY2584702.

ELIGIBILITY:
Inclusion Criteria:

Male participants:

• Agree to use a reliable method of birth control during the study and for at least 1 month following the last dose of study drug

Female participants:

• Women not of childbearing potential due to surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or menopause. Women with an intact uterus are deemed postmenopausal if they are greater than or equal to 45 years old, who have not taken hormones or oral contraceptives within the last year, and had cessation of menses for at least 1 year, or who have had 6 to 12 months of amenorrhea with follicle-stimulating hormone (FSH) levels consistent with postmenopausal state.

All participants:

* have a screening body mass index (BMI) of 18.5 to 32.0 kilograms per square meter (kg/m^2), inclusive
* have clinical laboratory test results within the normal range for the population or investigator site, or with abnormalities deemed clinically insignificant by the investigator. In particular, participants should have normal or near normal screening liver tests at the discretion of the investigator
* have normal blood pressure and pulse rate (supine) at screening, or with minor deviations judged to be acceptable by the investigator
* have venous access sufficient to allow blood sampling as per the protocol
* are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* have given written informed consent approved by Lilly and the ethical review board (ERB) governing the site

Exclusion Criteria

All participants:

* are currently enrolled in, have completed or discontinued within the last 30 days from, a clinical trial involving an investigational product other than the investigational product used in this study; or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study. Participants that participate in Part A of this study may participate in Part B of the study if the first dosing in Part B is >30 days after the dose of LY2584702 or placebo in Part A.
* have known allergies to LY2584702, or related compounds
* have an abnormality in the 12-lead electrocardiogram (ECG) [including but not limited to Bazett's corrected QT (QTcB) interval >450 milliseconds (msec) for men and >470 msec for women]
* have a history within the last 2 years or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* have a history of drug or alcohol abuse, or regularly use known drugs of abuse
* show evidence of human immunodeficiency virus infection and/or positive human immunodeficiency virus (HIV) antibodies
* show evidence of hepatitis B and/or positive hepatitis B surface antigen
* intend to use over-the-counter or prescription medication within 14 days prior to dosing or during the study
* use of herbal supplements, grapefruit juice, grapefruits, Seville orange juice, Seville oranges, or Starfruit within 7 days prior to study dosing or intended use during the study
* have donated blood of more than 450 milliliters (mL) within the last 3 months
* have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females), or are unwilling to stop alcohol consumption from prior to dosing until the completion of each study period [ unit = 12 ounces (oz) or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits]

Applicable for Part A only:

• have known allergies to lignocaine, adrenaline, tetracycline, or related compounds, which will be used in the skin biopsy procedure

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part A: single period, single dose pilot assessed safety, tolerability. Part B: 4-period crossover evaluated bioavailability of 2 drug formulations. Part B, Period (P) 4 participants (pts) separated into 2 cohorts, received drug under fed (P4a) or fasted (P4b) conditions. Pts who withdrew or were withdrawn prior to completing P3 were replaced.
Groups:
- LY2584702: Participants enrolled in Part A of the study received a single dose of 25 milligrams (mg) LY2584702 (LY) reference formulation [RF (capsule)] in a fasted state on Day 1.
- Placebo: Participants enrolled in Part A of the study received placebo in a fasted state on Day 1.
- 10 mg LY TF, Placebo, 50 mg LY TF, 50 mg LY TF Fed: Participants enrolled in Part B of the study received a single dose of 10 mg LY2584702 test formulation [TF (tablet)], placebo, and 50 mg LY2584702 TF in a fasted state, on Day 1 of Periods 1, 2, and 3, respectively and 50 mg LY2584702 TF in a fed state in Period 4a, Day 1. There was a washout of at least 3 days between periods.
- Placebo, 50 mg LY RF, 50 mg LY TF, 50 mg LY TF Fed: Participants enrolled in Part B of the study received a single dose of placebo, 50 mg LY2584702 RF, and 50 mg LY2584702 TF in a fasted state, on Day 1 of Periods 1, 2, and 3, respectively and 50 mg LY2584702 TF in a fed state in Period 4a, Day 1. There was a washout of at least 3 days between periods.
- Placebo, 50 mg LY RF, 50 mg LY TF, 200 mg LY TF Fasted: Participants enrolled in Part B of the study received a single dose of placebo, 50 mg LY2584702 RF, and 50 mg LY2584702 TF in a fasted state, on Day 1 of Periods 1, 2, and 3, respectively and 200 mg LY2584702 TF in a fasted state in Period 4b, Day 1. There was a washout of at least 3 days between periods.
- 10 mg LY TF, 50 mg LY RF, 50 mg LY TF, 50 mg LY TF Fed: Participants enrolled in Part B of the study received a single dose of 10 mg LY2584702 TF, 50 mg LY2584702 RF, and 50 mg LY2584702 TF in a fasted state, on Day 1 of Periods 1, 2, and 3, respectively and 50 mg LY2584702 TF in a fed state in Period 4a, Day 1. There was a washout of at least 3 days between periods.
- 10 mg LY TF, 50 mg LY RF, 50 mg LY TF, 200 mg LY TF Fasted: Participants enrolled in Part B of the study received a single dose of 10 mg LY2584702 TF, 50 mg LY2584702 RF, and 50 mg LY2584702 TF in a fasted state, on Day 1 of Periods 1, 2, and 3, respectively and 200 mg LY2584702 TF in a fasted state in Period 4b, Day 1. There was a washout of at least 3 days between periods.
- 10 mg LY TF, 50 mg LY RF, 50 mg LY TF, Placebo Fasted: Participants enrolled in Part B of the study received a single dose of 10 mg LY2584702 TF, 50 mg LY2584702 RF, and 50 mg LY2584702 TF in a fasted state, on Day 1 of Periods 1, 2, and 3, respectively and placebo in a fasted state in Period 4b, Day 1. There was a washout of at least 3 days between periods.
- 10 mg LY TF, 50 mg LY RF, Placebo, 200 mg LY TF Fasted: Participants enrolled in Part B of the study received a single dose of 10 mg LY2584702 TF, 50 mg LY2584702 RF, and placebo in a fasted state, on Day 1 of Periods 1, 2, and 3, respectively and 200 mg LY2584702 TF in a fasted state in Period 4b, Day 1. There was a washout of at least 3 days between periods.
- 200 mg LY TF Fasted: Participant enrolled in Part B, Period 4b of the study received a single dose of 200 mg LY2584702 TF in a fasted state on Day 1.
Period: First Intervention (Period 1)
Arm/Group | LY2584702 | Placebo | 10 mg LY TF, Placebo, 50 mg LY TF, 50 mg LY TF Fed | Placebo, 50 mg LY RF, 50 mg LY TF, 50 mg LY TF Fed | Placebo, 50 mg LY RF, 50 mg LY TF, 200 mg LY TF Fasted | 10 mg LY TF, 50 mg LY RF, 50 mg LY TF, 50 mg LY TF Fed | 10 mg LY TF, 50 mg LY RF, 50 mg LY TF, 200 mg LY TF Fasted | 10 mg LY TF, 50 mg LY RF, 50 mg LY TF, Placebo Fasted | 10 mg LY TF, 50 mg LY RF, Placebo, 200 mg LY TF Fasted | 200 mg LY TF Fasted
Started | 8 | 2 | 2 | 1 | 3 (Replacement participant repeated Periods 1, 2 to fulfill treatment arm comparison requirements.) | 5 | 3 | 1 | 1 | 0
Completed | 8 | 2 | 2 | 1 | 3 | 5 | 3 | 1 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 1
Arm/Group | LY2584702 | Placebo | 10 mg LY TF, Placebo, 50 mg LY TF, 50 mg LY TF Fed | Placebo, 50 mg LY RF, 50 mg LY TF, 50 mg LY TF Fed | Placebo, 50 mg LY RF, 50 mg LY TF, 200 mg LY TF Fasted | 10 mg LY TF, 50 mg LY RF, 50 mg LY TF, 50 mg LY TF Fed | 10 mg LY TF, 50 mg LY RF, 50 mg LY TF, 200 mg LY TF Fasted | 10 mg LY TF, 50 mg LY RF, 50 mg LY TF, Placebo Fasted | 10 mg LY TF, 50 mg LY RF, Placebo, 200 mg LY TF Fasted | 200 mg LY TF Fasted
Started | 0 (Pts completed one period and did not enter washout for Part A.) | 0 (Pts completed one period and did not enter washout for Part A.) | 2 | 1 | 3 | 5 | 3 | 1 | 1 | 0
Completed | 0 | 0 | 2 | 1 | 3 | 5 | 3 | 1 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (Period 2)
Arm/Group | LY2584702 | Placebo | 10 mg LY TF, Placebo, 50 mg LY TF, 50 mg LY TF Fed | Placebo, 50 mg LY RF, 50 mg LY TF, 50 mg LY TF Fed | Placebo, 50 mg LY RF, 50 mg LY TF, 200 mg LY TF Fasted | 10 mg LY TF, 50 mg LY RF, 50 mg LY TF, 50 mg LY TF Fed | 10 mg LY TF, 50 mg LY RF, 50 mg LY TF, 200 mg LY TF Fasted | 10 mg LY TF, 50 mg LY RF, 50 mg LY TF, Placebo Fasted | 10 mg LY TF, 50 mg LY RF, Placebo, 200 mg LY TF Fasted | 200 mg LY TF Fasted
Started | 0 | 0 | 2 | 1 | 3 | 5 | 3 | 1 | 1 | 0
Completed | 0 | 0 | 2 | 1 | 3 | 5 | 3 | 1 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2
Arm/Group | LY2584702 | Placebo | 10 mg LY TF, Placebo, 50 mg LY TF, 50 mg LY TF Fed | Placebo, 50 mg LY RF, 50 mg LY TF, 50 mg LY TF Fed | Placebo, 50 mg LY RF, 50 mg LY TF, 200 mg LY TF Fasted | 10 mg LY TF, 50 mg LY RF, 50 mg LY TF, 50 mg LY TF Fed | 10 mg LY TF, 50 mg LY RF, 50 mg LY TF, 200 mg LY TF Fasted | 10 mg LY TF, 50 mg LY RF, 50 mg LY TF, Placebo Fasted | 10 mg LY TF, 50 mg LY RF, Placebo, 200 mg LY TF Fasted | 200 mg LY TF Fasted
Started | 0 | 0 | 2 | 1 | 3 | 5 | 3 | 1 | 1 | 0
Completed | 0 | 0 | 2 | 1 | 2 (One participant discontinued Washout Period 2 and was replaced in Period 1.) | 5 | 3 | 1 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (Period 3)
Arm/Group | LY2584702 | Placebo | 10 mg LY TF, Placebo, 50 mg LY TF, 50 mg LY TF Fed | Placebo, 50 mg LY RF, 50 mg LY TF, 50 mg LY TF Fed | Placebo, 50 mg LY RF, 50 mg LY TF, 200 mg LY TF Fasted | 10 mg LY TF, 50 mg LY RF, 50 mg LY TF, 50 mg LY TF Fed | 10 mg LY TF, 50 mg LY RF, 50 mg LY TF, 200 mg LY TF Fasted | 10 mg LY TF, 50 mg LY RF, 50 mg LY TF, Placebo Fasted | 10 mg LY TF, 50 mg LY RF, Placebo, 200 mg LY TF Fasted | 200 mg LY TF Fasted
Started | 0 | 0 | 2 | 1 | 2 | 7 (Replacement pts repeated Period (P) 3 to fulfill requirement for P3 versus P4a comparison.) | 3 | 1 | 1 | 0
Completed | 0 | 0 | 2 | 1 | 2 | 7 | 3 | 1 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 3
Arm/Group | LY2584702 | Placebo | 10 mg LY TF, Placebo, 50 mg LY TF, 50 mg LY TF Fed | Placebo, 50 mg LY RF, 50 mg LY TF, 50 mg LY TF Fed | Placebo, 50 mg LY RF, 50 mg LY TF, 200 mg LY TF Fasted | 10 mg LY TF, 50 mg LY RF, 50 mg LY TF, 50 mg LY TF Fed | 10 mg LY TF, 50 mg LY RF, 50 mg LY TF, 200 mg LY TF Fasted | 10 mg LY TF, 50 mg LY RF, 50 mg LY TF, Placebo Fasted | 10 mg LY TF, 50 mg LY RF, Placebo, 200 mg LY TF Fasted | 200 mg LY TF Fasted
Started | 0 | 0 | 2 | 1 | 2 | 7 | 3 | 1 | 1 | 0
Completed | 0 | 0 | 2 | 1 | 2 | 5 (Two participants (pts) discontinued Washout P3 and were replaced in P3.) | 3 | 1 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Period: Forth Intervention (Period 4a/4b)
Arm/Group | LY2584702 | Placebo | 10 mg LY TF, Placebo, 50 mg LY TF, 50 mg LY TF Fed | Placebo, 50 mg LY RF, 50 mg LY TF, 50 mg LY TF Fed | Placebo, 50 mg LY RF, 50 mg LY TF, 200 mg LY TF Fasted | 10 mg LY TF, 50 mg LY RF, 50 mg LY TF, 50 mg LY TF Fed | 10 mg LY TF, 50 mg LY RF, 50 mg LY TF, 200 mg LY TF Fasted | 10 mg LY TF, 50 mg LY RF, 50 mg LY TF, Placebo Fasted | 10 mg LY TF, 50 mg LY RF, Placebo, 200 mg LY TF Fasted | 200 mg LY TF Fasted
Started | 0 | 0 | 2 | 1 | 2 | 5 | 3 | 1 | 1 | 1 (One pt was enrolled directly into P4b to fulfill requirement for safety and tolerability assessment.)
Completed | 0 | 0 | 2 | 1 | 2 | 5 | 3 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Part A (LY2584702): Participants enrolled in Part A of the study received a single dose of 25 milligrams (mg) LY2584702 (LY) reference formulation [RF (capsule)] in a fasted state on Day 1.
- Part A (Placebo): Participants enrolled in Part A of the study received placebo in a fasted state on Day 1.
- Total: Total of all reporting groups
Arm/Group | Part A (LY2584702) | Part A (Placebo) | 10 mg LY TF, Placebo, 50 mg LY TF, 50 mg LY TF Fed | Placebo, 50 mg LY RF, 50 mg LY TF, 50 mg LY TF Fed | Placebo, 50 mg LY RF, 50 mg LY TF, 200 mg LY TF Fasted | 10 mg LY TF, 50 mg LY RF, 50 mg LY TF, 50 mg LY TF Fed | 10 mg LY TF, 50 mg LY RF, 50 mg LY TF, 200 mg LY TF Fasted | 10 mg LY TF, 50 mg LY RF, 50 mg LY TF, Placebo Fasted | 10 mg LY TF, 50 mg LY RF, Placebo, 200 mg LY TF Fasted | 200 mg LY TF Fasted | Total
Number analyzed (Participants) | 8 | 2 | 2 | 1 | 3 | 7 | 3 | 1 | 1 | 1 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.9 (7.3) | 24 (4.2) | 44 (25.5) | 39 | 28 (8.2) | 34 (6.1) | 34 (8.9) | 28 | 35 | 28 | 32.6 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 8 | 2 | 2 | 1 | 3 | 7 | 3 | 1 | 1 | 1 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 8 | 2 | 2 | 1 | 3 | 7 | 3 | 1 | 1 | 1 | 29
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 8 | 2 | 2 | 1 | 3 | 7 | 3 | 1 | 1 | 1 | 29

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Maximum Observed Plasma Concentration (Cmax)
Description: The Cmax following a single oral dose of LY2584702 test formulation [TF (tablet)] or reference formulation [RF (capsule)] is reported.
Time Frame: Part A: Day 1 and Part B: Periods 1 to 4, Day 1 [Predose, 1 hour (h), 3 h, 4 h, 6 h, 10 h, 24 h, 48 h postdose]
Population: Randomized participants in Part A or B of the study who had evaluable Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- 25 mg LY2584702 RF Fasted: Participants received a 25 milligram (mg) LY2584702 RF orally in a fasted state on Day 1 in Part A of the study.
- 10 mg LY2584702 TF Fasted: Participants received 10 mg of LY2584702 TF orally in a fasted state, in Period 1, Day 1 of Part B of the study.
- 50 mg LY2584702 RF Fasted: Participants received 50 mg of LY2584702 RF orally in a fasted state, in Period 2, Day 1 of Part B of the study.
- 50 mg LY2584702 TF Fasted: Participants received 50 mg of LY2584702 TF orally in a fasted state, in Period 3, Day 1 of Part B of the study.
- 50 mg LY2584702 TF Fed: Participants received 50 mg of LY2584702 TF orally in a fed state, in Period 4a, Day 1 of Part B of the study.
- 200 mg LY2584702 TF Fasted: Participants received 200 mg of LY2584702 TF orally in a fasted state, in Period 4b, Day 1 of Part B of the study.
Arm/Group | 25 mg LY2584702 RF Fasted | 10 mg LY2584702 TF Fasted | 50 mg LY2584702 RF Fasted | 50 mg LY2584702 TF Fasted | 50 mg LY2584702 TF Fed | 200 mg LY2584702 TF Fasted
Number analyzed (Participants) | 8 | 12 | 14 | 16 | 8 | 7
nanograms per milliliter (ng/mL) | 266.83 (71) | 198.22 (26) | 481.11 (39) | 668.87 (26) | 794.13 (27) | 1486.5 (11)

2. Secondary Outcome: Pharmacokinetics, Area Under the Concentration-Time Curve (AUC)
Description: AUC from time 0 to the time of the last quantifiable concentration [AUC(0-tlast)] and AUC from time 0 to infinity [AUC(0-inf)] following a single oral dose of LY2584702 test formulation [TF (tablet)] or reference formulation [RF (capsule)] is reported.
Time Frame: Part A: Day 1 and Part B: Periods 1 to 4, Day 1 [Predose, 1 hour (h), 3 h, 4 h, 6 h, 10 h, 24 h, 48 h postdose]
Population: Randomized participants in Part A or B of the study who had evaluable AUC data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*h/mL)
Arm/Group | 25 mg LY2584702 RF Fasted | 10 mg LY2584702 TF Fasted | 50 mg LY2584702 RF Fasted | 50 mg LY2584702 TF Fasted | 50 mg LY2584702 TF Fed | 200 mg LY2584702 TF Fasted
Number analyzed (Participants) | 8 | 12 | 14 | 16 | 8 | 7
nanograms*hour per milliliter (ng*h/mL)
  AUC(0-tlast) | 1740 (63) | 1070 (26) | 3310 (43) | 4210 (25) | 5560 (30) | 10300 (20)
  AUC(0-inf) | 1860 (58) | 1110 (27) | 3530 (43) | 4430 (25) | 5620 (29) | 10900 (20)

3. Secondary Outcome: Part B: Baseline-Adjusted Change-From-Predose in the Concentration of Lipids (Total Cholesterol)
Description: Baseline-adjusted change-from-predose in lipid concentrations were measured to assess the LY2584702 effect on lipids under different fed states. The 50-milligram (mg) LY2584702 test formulation [TF (tablet)] was the only dose and formulation administered in both the fasted and fed states for comparison. Therefore, changes in total cholesterol after single oral doses of placebo, 10-mg, or 200-mg LY2584702 TF or 25-mg or 50-mg LY2584702 reference formulation [RF (capsule)] were not calculated. The baseline-adjusted change-from-predose in total cholesterol levels in the fasted and fed state following a single 50-mg LY2584702 TF dose is reported. Baseline was Day -1 of Period 1 for Period 3 fasted state and baseline was Day -1 of Period 4a for Period 4a fed state. Least squares (LS) means was calculated using mixed model repeating measures (MMRM) and adjusted for treatment, time, treatment by time, and participant.
Time Frame: Part B: Baseline [Periods 1 and 4a (Day -1)], Periods 3, 4a (Day 1). Lipid concentration measurements were performed at time point 0 and 1 hour (h), 3 h, 4 h, 6 h, 10 h, and 24 h.
Population: Randomized participants (pts) in Part B of study who had both baseline and postdose total cholesterol measurements. Pts not analyzed for baseline-adjusted change-from-predose total cholesterol levels after single dose placebo, 10-mg, or 200-mg LY2584702 TF or 25-mg or 50-mg LY2584702 RF since they weren't administered in both fasted and fed state.
Measure: Least Squares Mean (90% Confidence Interval); unit: milligrams per deciliter (mg/dL)
Arm/Group | 50 mg LY2584702 TF Fasted | 50 mg LY2584702 TF Fed
Number analyzed (Participants) | 13 | 8
milligrams per deciliter (mg/dL)
  1-hour postdose | -5.62 [-11.53 to 0.30] | -2.38 [-9.91 to 5.16]
  3-hours postdose | -4.00 [-9.91 to 1.91] | -1.75 [-9.29 to 5.79]
  4-hours postdose | -4.15 [-10.07 to 1.76] | -1.88 [-9.41 to 5.66]
  6-hours postdose | -4.77 [-10.68 to 1.14] | 0.75 [-6.79 to 8.29]
  10-hours postdose | -9.23 [-15.14 to -3.32] | -5.25 [-12.79 to 2.29]
  24-hours postdose | -8.85 [-14.76 to -2.93] | -8.75 [-16.29 to -1.21]

4. Secondary Outcome: Part A: QT Interval Corrected by Fridericia's Formula (QTcF) Change From Baseline to Day 1
Description: The QT interval is a measure of the time between the start of the Q wave and the end of the T wave and is calculated from electrocardiogram (ECG) data. Corrected QT (QTc) is the QT interval corrected for heart rate and RR, which is the interval between 2 R waves. Using Fridericia's formula: QTcF = QT/RR^0.33. The QTcF after single oral doses of LY2584702 reference formulation [RF (capsule)] were administered in a fasted state are reported at baseline (Day 1, Predose) and 3 hours (h), 4 h, 6 h, and 24 h postdose.
Time Frame: Part A: Baseline [Day 1 (Predose)] and Day 1 (3 h, 4 h, 6 h, and 24 h postdose)
Population: Randomized participants in Part A of the study who had both baseline and postdose ECG assessments at each time point. Data was not collected for Placebo group due to insufficient participants (N=2).
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Groups:
- 25 mg LY2584702 RF Fasted: Participants received a 25 milligram (mg) LY2584702 RF orally, in a fasted state on Day 1 in Part A of the study.
Arm/Group | 25 mg LY2584702 RF Fasted
Number analyzed (Participants) | 8
milliseconds (ms)
  Predose (Baseline) | 402.8 (14.4)
  3-hours postdose | 394.8 (12.6)
  4-hours postdose | 396.6 (10.7)
  6-hours postdose | 395.7 (12.8)
  24-hours postdose | 396.1 (10.6)

5. Secondary Outcome: Part B: Average Time-Matched QT Interval Corrected by Fridericia's Formula (QTcF) Change From Baseline to Day 1
Description: The QT interval is a measure of the time between the start of the Q wave and the end of the T wave and is calculated from electrocardiogram (ECG) data. Corrected QT (QTc) is the QT interval corrected for heart rate and RR, which is the interval between 2 R waves. Using Fridericia's formula: QTcF = QT/RR^0.33. The QTcF after single oral doses of LY2584702 test formulation [TF (tablet)], LY2584702 reference formulation [RF (capsule)], or placebo were administered in a fasted or fed state are reported at baseline (time-matched Day -1 QTcF) and 3 hours (h), 4 h, 6 h, and 24 h postdose. Day 1, Hour 24 was time-matched with Day-1, Hour 0.
Time Frame: Part B: Baseline [Period 1 (Day -1)] and Periods 1 to 4 (Day 1). Electrocardiograms (ECG) were performed at time point 0 and 3 h, 4 h, 6 h, and 24 h.
Population: Randomized participants in Part B of the study who had both baseline and postdose ECG assessments at each time point.
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Groups:
- 10 mg LY2584702 TF Fasted: Participants received 10 milligrams (mg) of LY2584702 TF orally in a fasted state in Period 1, Day 1 of Part B of the study.
- 50 mg LY2584702 RF Fasted: Participants received 50 mg of LY2584702 RF orally in a fasted state in Period 2, Day 1 of Part B of the study.
- 50 mg LY2584702 TF Fasted: Participants received 50 mg of LY2584702 TF orally in a fasted state in Period 3, Day 1 of Part B of the study.
- 50 mg LY2584702 TF Fed: Participants received 50 mg of LY2584702 TF orally in a fed state in Period 4a, Day 1 of Part B of the study.
- 200 mg LY2584702 TF Fasted: Participants received 200 mg of LY2584702 TF orally in a fasted state in Period 4b, Day 1 of Part B of the study.
- Placebo (Part B): Participants received placebo orally in a fasted state, in Periods 1 to 4, Day 1 of Part B of the study.
Arm/Group | 10 mg LY2584702 TF Fasted | 50 mg LY2584702 RF Fasted | 50 mg LY2584702 TF Fasted | 50 mg LY2584702 TF Fed | 200 mg LY2584702 TF Fasted | Placebo (Part B)
Number analyzed (Participants) | 12 | 14 | 16 | 8 | 7 | 8
milliseconds (ms)
  Day-1, Hour 0 (time-matched baseline) | 419.1 (21.0) | 413.6 (21.5) | 417.1 (18.9) | 428.0 (11.2) | 415.8 (23.5) | 416.4 (19.2)
  Day 1, Hour 0 | 416.4 (17.8) | 413.3 (23.0) | 414.4 (17.7) | 407.8 (16.2) | 413.1 (22.1) | 412.1 (19.8)
  Day-1, Hour 3 (time-matched baseline) | 416.1 (21.0) | 412.4 (19.8) | 413.8 (18.2) | 423.3 (14.8) | 415.2 (22.0) | 415.7 (14.2)
  Day 1, Hour 3 | 413.6 (17.8) | 410.6 (23.2) | 409.2 (16.2) | 402.6 (10.0) | 409.9 (22.1) | 412.3 (17.8)
  Day-1, Hour 4 (time-matched baseline) | 415.5 (20.6) | 413.1 (20.7) | 414.6 (18.3) | 420.7 (10.1) | 418.3 (24.2) | 413.4 (17.1)
  Day 1, Hour 4 | 414.8 (17.7) | 412.0 (21.0) | 409.2 (14.0) | 407.3 (12.1) | 413.3 (20.4) | 415.2 (19.3)
  Day-1, Hour 6 (time-matched baseline) | 417.1 (20.6) | 415.0 (19.8) | 417.6 (19.3) | 420.5 (12.5) | 422.3 (24.0) | 418.1 (16.8)
  Day 1, Hour 6 | 413.2 (14.8) | 410.6 (18.1) | 409.6 (14.3) | 414.8 (11.5) | 415.6 (15.8) | 412.4 (16.6)
  Day 1, Hour 24 | 415.4 (19.4) | 408.9 (19.0) | 409.1 (13.9) | 411.1 (13.5) | 409.0 (17.9) | 409.0 (19.8)

ADVERSE EVENTS:
Groups:
- Placebo: Participants received placebo orally in fasted state on Day 1 in Part A and Periods 1 to 4, Day 1 in Part B of the study.
- 25 mg LY2584702 RF Fasted: Participants received a 25 milligram (mg) LY2584702 reference formulation [RF (capsule)] orally in a fasted state on Day 1 in Part A of the study.
- 10 mg LY2584702 TF Fasted: Participants received 10 mg of LY2584702 test formulation [TF (tablet)] orally in a fasted state, in Period 1, Day 1 of Part B of the study.
Arm/Group | Placebo | 25 mg LY2584702 RF Fasted | 10 mg LY2584702 TF Fasted | 50 mg LY2584702 RF Fasted | 50 mg LY2584702 TF Fasted | 50 mg LY2584702 TF Fed | 200 mg LY2584702 TF Fasted
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8 | 0/12 | 0/14 | 0/16 | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 4/10 | 6/8 | 5/12 | 3/14 | 2/16 | 4/8 | 4/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | 25 mg LY2584702 RF Fasted (N=8) | 10 mg LY2584702 TF Fasted (N=12) | 50 mg LY2584702 RF Fasted (N=14) | 50 mg LY2584702 TF Fasted (N=16) | 50 mg LY2584702 TF Fed (N=8) | 200 mg LY2584702 TF Fasted (N=7)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site haematoma (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site related reaction (General disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 2 (3) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural site reaction (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes